CLINICAL TRIAL: NCT03247855
Title: Safety and Efficacy of Multivessel Minimally Invasive Coronary Artery Bypass Graft Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mohammed Farouk Abdel Hafez (Other)
Responsible Party: Sponsor-Investigator, Mohammed Farouk Abdel Hafez, assistant lecturer, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17200098
Record Dates: First submitted 2017-07-30; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimal invasive coronary artery bypass graft (Other)
  Interventions: Procedure: minimal invasive coronary artery bypass graft surgery

INTERVENTIONS:
Procedure: minimal invasive coronary artery bypass graft surgery — coronary artery bypass grafting surgery by using a minimal invasive technique

SUMMARY:
the aim of this study is to evaluate safety and efficacy of multivessel minimally invasive coronary artery bypass graft surgery through evaluating the possibility of reaching complete revascularization , the complications during surgery and the outcomes

DETAILED DESCRIPTION:
Minimally invasive direct coronary artery bypass (MIDCAB) grafting can achieve adequate coronary artery revascularization in a less invasive manner than conventional coronary artery bypass grafting (CABG). Bypass from the internal mammary artery (IMA) to the left anterior descending coronary artery (LAD) is an effective technique for the treatment of simple anterior descending artery disease. This surgery is especially recommended for patients with multiple lesions that are not suitable for stent stenosis . One of the main advantages of MIDCAB is that there is no need for cardiac arrest and cardiopulmonary bypass (CPB) transfer during surgery . MIDCAB patients also benefit from the neurological protection associated with this minimally invasive procedure . Unlike traditional revascularization techniques, which are highly invasive due to the use of a large incision (sternotomy) and cardiopulmonary bypass (CPB), MIDCAB limits invasiveness by operating through a small incision (thoracotomy) and by operating on the beating heart to avoid the need for CPB . By limiting invasiveness in these ways, MIDCAB can reduce the risk of complications such as infection and stroke . In comparison to traditional CABG and off-pump CABG (via a sternotomy), MIDCAB can enhance early post-operative quality of life and recovery time . Minimally invasive multivessel coronary surgery-coronary artery bypass grafting (MICS-CABG) through a small thoracotomy has many advantages over minimally invasive direct coronary artery bypass (MIDCAB). First, MIDCAB is limited to a single anastomosis of the left internal mammary artery to the left anterior descending artery (LIMA-LAD). The surgical exposure of MICS-CABG is done more laterally, leading to reduced risk of costochondral or rib injury. Also, MICS-CABG allows revascularization with a similar configuration to that of a traditional sternotomy technique, by direct-vision LIMA harvesting and hand-sewn proximal and distal anastomoses . MICS may be performed with or without cardiopulmonary bypass (CPB) assistance, but the use of femorofemoral CPB in multivessel revascularization has shown to be safe, mitigate the learning curve, prevent conversions, and allows operative time like that of a sternotomy. ]. Other advantages include a diminished need for blood transfusion, decreased surgical site infection rates, also early return to full physical function .

On the other hand complications include sternotomy conversion and development of left-sided pleural effusion . Postoperative pain can be an issue early, but it is transient, controllable, and significantly decreased by the third postoperative day; it is also associated with an overall improved postoperative pain picture with improved pulmonary functions . However, unlike sternotomy patients, MICS-CABG patients have no physical restriction postoperatively, which leads to better independence.

This study aim to evaluate Safety and efficacy of multivessel minimally invasive coronary artery bypass graft surgery through measuring several factors such as

1. measuring rate of intraoperative complications occurrence
2. measuring rate of intraoperative conversion to open sternotomy
3. measuring amount of post operative bleeding
4. measuring post operative pain
5. measuring rate of reexploration
6. measuring rate of wound infection
7. calculating days of postoperative hospital stay
8. calculating time to regain normal activity

The information gathered from the eligible patients will be entered into a data sheet containing the variables of interest that will be analyzed later at the end of the study. This study will not alter the patients' treatment and follow up at our center, by any means.

The following variables will be studied whenever applicable and whenever they are available in the patients' charts:

1. Demographic data: (Medical Record Number ,Sex ,Age Other comorbidity)
2. Preoperative variables : (chest pain , dyspnea ,ECG findings ,Myocardial markers and cardiac troponin ,Cardiac Angiography )
3. Operative variables: (Conversion to sternotomy. , Cardiac arrest ,Operation time ,Need for IABP, CPB ,Need for blood transfusion)
4. Postoperative variables: (Mortality , Bleeding , Pain , Need of reexploration , Hospital stay , Wound infection , Regain of normal activity , Relief of symptoms , Need for another revascularization within 6 month)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or more
2. Angiographically Indication for revascularization based upon symptoms of angina and/or objective evidence of myocardial ischemia
3. Suitable minimally invasive coronary surgery (MICS) candidate for non-emergent first time, single or multivessel coronary artery bypass grafting (on pump or off pump)
4. Willing and able to provide written informed consent and comply with study requirements and accepting the need of conversion if needed.
5. Patient is willing to comply with all follow-up visits

Exclusion Criteria:

1. Severe congestive heart failure (class III or IV according to NYHA, or pulmonary edema, cardiogenic shock) at the time of enrollment.
2. Prior surgery with the opening of pericardium or pleura.
3. Prior stroke (within 6 months)or more than 6 months if there are substantial neurological defects.
4. Acute ST-elevation MI within 72 hours prior to enrollment requiring revascularization.
5. Planned simultaneous surgical procedure unrelated to coronary revascularization (e.g. valve repair/replacement, aneurysmectomy, carotid endarterectomy or carotid stenting).
6. Contraindication to either CABG, MIDCAB or PCI/DES because of a coexisting clinical condition.
7. Significant leukopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis.
8. Intolerance or contraindication to aspirin or both clopidogrel and ticlopidine
9. Extra-cardiac illness that is expected to limit survival to less than 5 years e.g. oxygen-dependent chronic obstructive pulmonary disease, active hepatitis or significant hepatic failure, severe renal disease.
10. Suspected pregnancy. A pregnancy test will be administered prerandomization to all women of child-bearing age.
11. Patient inaccessible for follow-up visits required by protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
measuring rate of intraoperative complications occurrence | 2 years
  measuring the rate of complications as bleeding , failure of complete revascularization and cardiac arrest during operation
measuring rate of intraoperative conversion to open sternotomy | 2 years
measuring amount of post operative bleeding | 2 years
  measuring the amount of bleeding in the drains in 48 hours post operative in cc
measuring post operative pain | 2 years
  measuring pain using wong-baker faces pain rating scale
measuring rate of reexploration | 2 years
  measuring the need of reexploration of the patient due to post operative massive bleeding
measuring rate of wound infection | 2 years
calculating days of postoperative hospital stay | 2 years
calculating time to regain normal activity | 2 years